CLINICAL TRIAL: NCT07227532
Title: Assessment of Long-Term Safety and Effectiveness in Treatment Management of Atrial Fibrillation With the VARIPULSE™ Catheter System
Brief Title: A Study Assessing Long-Term Safety and Effectiveness in Treatment Management of Atrial Fibrillation With VARIPULSE Catheter System
Acronym: AdmIREPAS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Biosense Webster, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BWI202405; BWI202405 (Other: Biosense Webster, Inc.)
Record Dates: First submitted 2025-11-11; First posted 2025-11-12 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Pulsed Field Ablation by VARIPULSE Catheter with TRUPULSE Generator (Experimental): Participants undergoing electrophysiology mapping and pulsed field ablation (PFA) for management of treatment of symptomatic paroxysmal atrial fibrillation (AF) will undergo pulmonary vein (PV) ablation with the VARIPULSE Catheter with a TRUPULSE Generator.
  Interventions: Device: Pulsed Field Ablation by VARIPULSE Catheter with TRUPULSE Generator

INTERVENTIONS:
Device: Pulsed Field Ablation by VARIPULSE Catheter with TRUPULSE Generator — Pulsed field ablation by VARIPULSE catheter with TRUPULSE generator will be used.

SUMMARY:
The purpose of this study is to evaluate the long-term safety and effectiveness of the VARIPULSE catheter system for pulmonary vein isolation (PVI) in the treatment of participants with symptomatic paroxysmal atrial fibrillation (PAF).

ELIGIBILITY:
Inclusion Criteria:

* Symptomatic paroxysmal Atrial Fibrillation (AF) who, in the opinion of the investigator, are candidates for catheter ablation for AF
* Refractory, intolerant, or contraindicated to Class I/III antiarrhythmic drugs (AAD)
* Willing and capable of providing consent
* Able and willing to comply with all pre-, post-, and follow-up testing and requirements

Exclusion Criteria:

* Previously diagnosed with persistent or long-standing persistent AF (more than [>] 7 days in duration)
* Previous surgical or catheter ablation for AF
* Significant congenital anomaly or medical problem that in the opinion of the investigator would be a contraindication to catheter ablation for AF
* Current enrollment in an investigational study evaluating another device or drug
* Life expectancy less than 12 months
* Any contraindications as defined in the Protocol

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 276 (Estimated)
Dates: Start 2025-10-21 (Actual); Primary Completion 2030-12-31 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
Occurences of Early Onset Primary Adverse Events (PAEs) Within 7 days of the Index Ablation Procedure | Within 7 days post index procedure
  PAE's will include the following adverse events: atrio-esophageal fistula, phrenic nerve paralysis, cardiac tamponade/perforation, pulmonary vein stenosis (PVS), device or procedure related death, stroke/cerebrovascular accident (CVA), major vascular access complication/bleeding, thromboembolism, myocardial infarction, transient ischemic attack (TIA), pericarditis, heart block, pulmonary edema (respiratory insufficiency), and vagal nerve injury/gastroparesis.
Freedom From Documented (Symptomatic and Asymptomatic) Atrial Tachyarrhythmias Episodes | Day 61-1095 post-index procedure
  Freedom from documented (symptomatic and asymptomatic) atrial tachyarrhythmias (atrial fibrillation [AF], atrial tachycardia [AT] or atrial flutter [AFL] of unknown origin) episodes will be reported. AFL of unknown origin is defined as all AFL except those Cavotricuspid isthmus CTI dependent AFL as confirmed by 12-Lead electrocardiogram (ECG) and entrainment maneuvers in an evaluation period study.

CONTACTS AND LOCATIONS:
Overall Officials: Biosense Webster, Inc. Clinical Trial, Study Director — Biosense Webster, Inc.
Locations (2):
- United States (2):
  - Community Memorial Hospital, Ventura, California
  - Mercy Hospital, Janesville, Wisconsin

IPD SHARING:
Plan to Share IPD: Yes
The data sharing policy of Johnson & Johnson Innovative Medicine is available at innovativemedicine.jnj.com/our-innovation/clinical-trials/transparency. As noted on this site, requests for access to the study data can be submitted through Yale Open Data Access (YODA) Project site at yoda.yale.edu
URL: https://innovativemedicine.jnj.com/our-innovation/clinical-trials/transparency